CLINICAL TRIAL: NCT03159533
Title: Project IMPACT: Community Health Care Worker (CHW) Intervention
Brief Title: Project IMPACT: CHW Intervention
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-00969
Record Dates: First submitted 2017-04-13; First posted 2017-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Step wedge design, whereby 5 groups of 3 practices will implement the intervention in phases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHW Intervention (Active Comparator): CHW lead Sessions Session1: BP and the Cardiovascular System Session 2: Nutrition and food labels Session 3: Physical Activity and Stress Management Session 4: CVD Risk factors: cholesterol, blood sugar, & Smoking Session 5: Health Communication, Healthcare access & Review
  Interventions: Behavioral: CHW Intervention
- Control Group (Placebo Comparator): Wait-list
  Interventions: Behavioral: Wait List Control Group

INTERVENTIONS:
Behavioral: CHW Intervention — Patients randomized to Group A will be invited to attend 4 more group educational sessions on self-management immediately.CHWs will follow up with participants by phone or in person through a home or clinic visit. At these follow-up meetings, CHWs will engage in goal-setting activities regarding changes to health behaviors, medication adherence, or other issues related to hypertension control as identified jointly by the patient and CHW. CHWs will also collect height, weight, and blood pressure measurements at initial and in-person follow-up visits. The CHW will make necessary referrals to other services available in the community (i.e. exercise classes, social services, mental health, tobacco cessation, etc.).
  Arms: CHW Intervention
Behavioral: Wait List Control Group — 4 education sessions beginning 6-12 months later.
  Arms: Control Group

SUMMARY:
The proposed study "Project IMPACT: CHW Intervention" is part of a larger study examining the efficacy, adoption, and impact of integrated EHR-based decision-support and physician feedback interventions with community health worker (CHW)-led self-management and coaching support for South Asian patients with uncontrolled hypertension. This is a randomized control intervention utilizing community health worker (CHW)-led self-management and coaching support for South Asian patients with uncontrolled hypertension at PCP clinics in New York City.

DETAILED DESCRIPTION:
The Goal of this study is that:

1. EHR-based decision support and performance feedback interventions will be more effective in improving hypertension control for South Asian patients than standard care;
2. A combined EHR-CHW intervention will be more effective in improving hypertension control for South Asian patients compared to standard care and the EHR-based intervention

Investigators hope to implement and assess the efficacy of CHW-led coaching through promotion of team-based care and use of culturally tailored education to improve hypertension control and mitigate risk factors related to CVD among South Asian patients with uncontrolled hypertension. Study findings can provide translatable and scalable models for other limited English proficient communities.

ELIGIBILITY:
Inclusion Criteria:

CHW Intervention

* Diagnosis of hypertension or at least two systolic blood pressure measurements of 140 mm Hg or greater, or at least two diastolic BP 90 mm Hg or greater in the past 12 months.

Focus Group

* Any clinical patients meeting the inclusion criteria for the CHW Intervention who participated in the CHW Intervention Pilot Round.

Exclusion Criteria:

* Pregnant patients are excluded.
* No children or vulnerable subjects will be enrolled in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Percent of current diagnosed hypertensive patients with BP <140/90 (or BP<130/80 for patients with diabetes) at 6 Months | 6 Months
Percent of current diagnosed hypertensive patients with BP <140/90 (or BP<130/80 for patients with diabetes) at 12 months | 12 months
Percent of patients with HbA1c <7 (for patients with hypertension + diabetes) at 6 months | 6 months

SECONDARY OUTCOMES:
Percent of patients with diagnosis of hypertension with a BP measure taken in the past 6 months | 6 months
Percent of patients without hypertension having valid BP measurement, last 12 months | 12 months
Percent of current hypertensive patients screened for diabetes in last year | 12 months
Percent of current hypertensive patients receiving counseling on BMI, diet and physical activity | 12 months
Percent of current diagnosed hypertensive patients referred to a nutritionist in the past year | 12 months
Percent of current diagnosed hypertensive patients who smoke who have been referred for smoking cessation | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Islam, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Islam NS, Wyatt LC, Ali SH, Zanowiak JM, Mohaimin S, Goldfeld K, Lopez P, Kumar R, Beane S, Thorpe LE, Trinh-Shevrin C. Integrating Community Health Workers into Community-Based Primary Care Practice Settings to Improve Blood Pressure Control Among South Asian Immigrants in New York City: Results from a Randomized Control Trial. Circ Cardiovasc Qual Outcomes. 2023 Mar;16(3):e009321. doi: 10.1161/CIRCOUTCOMES.122.009321. Epub 2023 Feb 23. PMID 36815464
- [Derived] Lopez PM, Zanowiak J, Goldfeld K, Wyka K, Masoud A, Beane S, Kumar R, Laughlin P, Trinh-Shevrin C, Thorpe L, Islam N. Protocol for project IMPACT (improving millions hearts for provider and community transformation): a quasi-experimental evaluation of an integrated electronic health record and community health worker intervention study to improve hypertension management among South Asian patients. BMC Health Serv Res. 2017 Dec 6;17(1):810. doi: 10.1186/s12913-017-2767-1. PMID 29207983